CLINICAL TRIAL: NCT02135198
Title: A Phase I Single Site, Single Dose, Randomised, Double-blind, Placebo Controlled 3-way Cross-over Biomarker Study Investigating the Effect of the GABA Modulator AZD7325 on Short Interval Intracortical Inhibition (SICI) in Healthy Volunteers
Brief Title: Effects of GABA Modulator AZD7325 on Cortical Excitability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 13/0231; 2013-005472-17 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-05-09 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: GABA modulator; AZD7325; Short interval intracortical inhibition; volunteers
MeSH Terms: interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 mg AZD7325 (Experimental): 2 mg AZD7325 in orange capsule, Size 0, single oral dose
  Interventions: Drug: 2 mg AZD7325; Drug: 10 mg AZD7325; Drug: Placebo
- 10 mg AZD7325 (Experimental): 10 mg AZD7325 in orange capsule, Size 0, singe oral dose
  Interventions: Drug: 2 mg AZD7325; Drug: 10 mg AZD7325; Drug: Placebo
- Placebo (Placebo Comparator): 10 mg Microcrystalline cellulose in orange capsule, Size 0, single oral dose
  Interventions: Drug: 2 mg AZD7325; Drug: 10 mg AZD7325; Drug: Placebo

INTERVENTIONS:
Drug: 2 mg AZD7325 — A single 2 mg oral dose of AZD7325
Drug: 10 mg AZD7325 — A single 10 mg oral dose of AZD7325
Drug: Placebo — A single oral dose

SUMMARY:
GABA (gamma-aminobutyric acid) is the main inhibitory compound in the human brain. Drugs that enhance its effects by binding on GABA receptors (e.g., benzodiazepines) are used to treat various diseases such as epilepsy, insomnia, anxiety or movement disorders. However, the use of these medications is often compromised due to their side effects, like sedation, cognitive impairment, and addiction.

Many of these side effects have been linked to a particular type of GABA receptor (GABA A alpha 1). Therefore, effort is being made to develop drugs that do not act on this receptor, but maintain their beneficial properties by acting on other types of GABA receptors. AZD7325 is a drug that selectively acts on GABA A alpha 2 and A alpha 3 receptors, but not A alpha 1. It has been tested in more than 700 people and so far proved to be generally well tolerated. Positron emission tomography (PET) study in humans demonstrated that AZD7325 binds to GABA A receptors in the brain after a single dose. Early clinical studies have shown that it has less sedative and cognitive adverse events as compared with a benzodiazepine lorazepam.

In this study, we will investigate its effects on short interval intracortical inhibition (SICI). SICI is neurophysiological marker of inhibitory processes in the motor cortex. It is obtained non-invasively by using transcranial magnetic stimulation (TMS). In TMS, magnetic impulses applied over the scalp that in turn induce a current in a small area of the brain. If applied over the motor areas of the brain, impulses result in muscle twitch that is recorded with surface electrodes. SICI is enhanced by certain drugs like benzodiazepines that act on GABA A alpha 1,2,3, and 5 receptor subtypes, but not by zolpidem acting solely on alpha 1 subtype. Because GABA A alpha 5 receptor subtype is less common in the cortex, it has been concluded that the drug effects on SICI are related to GABA A alpha 2 and alpha 3 receptors.

If AZD7325 proves to enhance SICI in healthy volunteers, this would create the grounds for the use of this medication to treat certain neurological disorders in which SICI has been found to be impaired (e.g., dystonia).

ELIGIBILITY:
Inclusion Criteria:

* Male adults aged 18 to 55 years (extremes are included)
* A body weight resulting in a body mass index (BMI) of 18 - 30 kg/m2 (extremes included) using the formula BMI = body-weight [in kg] / body-height [in m]2
* Able and willing to sign the Informed Consent Form prior to screening evaluations
* History of good physical and mental health as determined by history taking and laboratory examinations, ECG, blood pressure and heart rate recordings as judged by the investigator
* Willing not to consume alcohol or to smoke or chew tobacco on days of assessments
* Subjects must be willing to avoid unprotected sex or donating sperm until 3 weeks after drug administration

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to AZD7325 or chemically related compounds or excipients which may be employed in the study or to any other drug used in the past
* Subject has taken systemically any potent or moderate CYP3A4 or CYP2C9 inhibitor, 1 month prior to screening (topical or inhaled are permitted) such as: aprepitant, barbiturates, carbamazepine, clarithromycin, erythromycin, cyclosporine, diltiazem, efavirenz, fluconazole, HIV protease inhibitors, glucocorticoids, itraconazole (oral/IV), ketoconazole, nefazodone, nevirapine, phenytoin, pioglitazone, primidone, rifabutin, rifampicin, telithromycin, St. John's wort, verapamil
* Use of any prescription drug within two weeks prior to the first dosing, except for topical medication without systemic exposure
* Clinically relevant history or presence of any medical disorder, potentially interfering with this trial
* Clinically relevant abnormal laboratory, ECG, HR or BP at screening as judged by the investigator
* History of or current abuse of drugs (including prescription medication) or alcohol or solvents
* Smoking in excess of 5 cigarettes per day or the equivalent within 28 days prior to the first study day
* Smoking or chewing of tobacco or consuming of alcohol 24 hours before and on the days of assessment
* Subject is family member or in the employment line management of study personnel
* Subject's partner is planning pregnancy within 3 months of last dosing
* Participation in an investigational medicinal product (IMP) intervention trial within last month or more than four in the previous 12 months
* Abnormal SICI response, kinematic analysis of circle drawing, SDMT, VAS outside 95% confidence interval of normal at screening visit
* Contraindications for TMS

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in conventional measure of percentage short interval intracortical inhibition (SICI) at an interstimulus interval (ISI) of 2.5 ms and conditioning stimulus intensity of 70 percent of resting motor threshold | baseline at 1, 2, and 8 hours after the study medication.

SECONDARY OUTCOMES:
Change in the variables of kinematic analysis of circle drawing | baseline at 1, 2, and 8 hours after the study medication
Change in the rating on a 0-100 mm Visual Analogue Scale (VAS) of degree of sedation and the score of Symbol Digit Modalities Test (SDMT) | baseline at 1, 2, and 8 hours after the study medication
Safety and tolerability of a single dose of AZD7325 by assessment of adverse events, vital signs, physical examination, ECG, and laboratory variables | 4 times ( before each dose and 48-96 hours after the last dose of study medication). Adverse events also at follow-up telephone call within a week after the last dose of study medication

OTHER OUTCOMES:
The change in the area under the curve of short interval intracortical inhibition (SICI) slope recruitment using conditioning stimulus intensities of 50, 60, 70, and 80 percent of resting motor threshold | baseline at 1, 2, and 8 hours after the study medication

CONTACTS AND LOCATIONS:
Overall Officials: Martin Koltzenburg, Prof, Principal Investigator — Institute of Neurology, University College London
Locations (1):
- National Hospital for Neurology and Neurosurgery, UCLH NHS Foundation Trust, London, United Kingdom